CLINICAL TRIAL: NCT05174351
Title: Effect of Beta-blocker Discontinuation on Functional Capacity and Cardiac Hemodynamics in Patients With Heart Failure With Preserved Ejection Fraction
Brief Title: Beta-blocker Discontinuation in Heart Failure With Preserved Ejection Fraction
Acronym: HFpEF-BB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Responsible Party: Principal Investigator, Christopher Pickett, Associate Professor, UConn Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-145-2
Record Dates: First submitted 2021-12-02; First posted 2021-12-30 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-07

CONDITIONS: Heart Failure With Preserved Ejection Fraction
Keywords: HFpEF; Beta-blocker; echocardiogram; 6MWT

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HFpEF patients (Experimental): HFpEF patient who are currently taking beta blockers
  Interventions: Other: beta blocker discontinuation

INTERVENTIONS:
Other: beta blocker discontinuation — beta blocker discontinuation

SUMMARY:
This is a prospective pilot study to evaluate changes before and 4 weeks after beta-blocker withdrawal in 30 HFpEF patients.

DETAILED DESCRIPTION:
This is a prospective pilot study to evaluate changes before and 4 weeks(+/- 1 week) after beta-blocker withdrawal in 30 HFpEF patients. The study involves 2 visits that are 4 weeks apart. The first study visit will occur at a standard of care clinic visit and the second visit will be a research visit to fill out questionnaires and perform the limited echocardiogram. No long term follow up beyond the 2nd visit.

ELIGIBILITY:
Inclusion Criteria:

* Stable HFpEF patients with NYHA Class II-III or elevated BNP ≥100
* N=30 (Target: 30).
* Age: 50 ~ 80 years.
* ECHO evidence of EF ≥50% and Grade 2 or 3 diastolic dysfunction.
* Chronic loop diuretic use
* Currently on beta-blocker

Exclusion Criteria:

* Beta blocker was prescribed for treating other cardiac conditions such as atrial fibrillation or coronary artery disease.
* Heart rate > 100 bpm
* Recent hospitalization due to HF within 3 months
* Non-English speaker

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-12-20 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Changes in KCCQ-23 score | Baseline and after 4 weeks of beta blocker discontinuation
  Kansa city cardiomyopathy questionnaire (KCCQ-23)- self-administered, 23-item. questionnaire that quantifies physical limitations, symptoms, self-efficacy, social interference and quality of life. Scores are transformed to a range of 0-100, where higher scores reflect better health status.

SECONDARY OUTCOMES:
Changes in cardiac mechanics by echocardiography | Baseline and after 4 weeks of beta blocker discontinuation
  Echocardiographic E/e' ratio
Changes in biomarker | Baseline and after 4 weeks of beta blocker discontinuation
  changes from baseline in BNP level (pg/mL) after 4 weeks of beta blocker discontinuation
6 minute walk test | Baseline and after 4 weeks of beta blocker discontinuation
  The distance (meters) covered over a time of 6 minutes. A greater distance indicates a better exercise capacity.

CONTACTS AND LOCATIONS:
Overall Officials: Kai Chen, MD,PhD, Principal Investigator — UConn Health
Locations (1):
- UConn Health / John Dempsey Hospital, Farmington, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No